CLINICAL TRIAL: NCT03015090
Title: Association Study Between CYP1A2 Gene Polymorphisms and Metabolism of Theophylline in Han and Uygur Patients With COPD
Brief Title: Association Study Between CYP1A2 Gene Polymorphisms and Metabolism of Theophylline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: XiaoGuang Zou (Other)
Collaborators: Southern Medical University, China (Other)
Responsible Party: Sponsor-Investigator, XiaoGuang Zou, Professor of Pharmacy, Kashgar 1st People's Hospital
Organization: Kashgar 1st People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016D01C013
Record Dates: First submitted 2017-01-03; First posted 2017-01-09 (Estimated); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; CYP1A2; Theophylline
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Theophylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- theophylline (Experimental)
  Interventions: Drug: Theophylline

INTERVENTIONS:
Drug: Theophylline — After oral theophylline 200mg per day for one week, blood sample will be collected for determining plasma concentrations of theophylline and it's metabolites and the genotypes of CYP1A2

SUMMARY:
The aim of this study is to determine whether common CYP1A2 gene polymorphisms effect metabolism of theophylline in Han and Uygur Patients with chronic obstructive pulmonary disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years,Weight 40-80kg COPD patients, male or female; regularly visiting our hospital; taking a sustained-release preparation of theophylline continuously for at least 2 weeks

Exclusion Criteria:

* Patients with renal or hepatic dysfunction; Patients with congestive heart failure; Patients with hypothyroidism or hyperthyroidism; Patients currently taking drugs likely to effect theophylline metabolism or who had taken such drugs in the preceding week; Patients with extreme obesity Patients with very severe Chronic Obstructive Pulmonary Disease(COPD)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of theophylline | one week
  Blood samples will be taken after receiving oral theophylline

CONTACTS AND LOCATIONS:
Locations (1):
- Kashgar 1st People's Hospital, Kashgar, Xinjiang, China

IPD SHARING:
Plan to Share IPD: Yes